CLINICAL TRIAL: NCT01769222
Title: A Phase I/II Study of Intratumoral Injection of Ipilimumab in Combination With Local Radiation in Melanoma, Non-Hodkgkin Lymphoma and Colorectal Carcinoma
Brief Title: Ipilimumab and Local Radiation for Selected Solid Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Planned Future Study
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, George Albert Fisher, Professor of Medicine, Stanford University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-25597; NCI-2012-02988 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); VAR0090 (Other: OnCore); 5136 (Other: Stanford IRB alternate)
Record Dates: First submitted 2013-01-14; First posted 2013-01-16 (Estimated); Results first posted 2017-03-03 (Actual); Last update posted 2024-01-24 (Actual); Status verified 2024-01

CONDITIONS: Adult Nasal Type Extranodal NK/T-cell Lymphoma; Anaplastic Large Cell Lymphoma; Angioimmunoblastic T-cell Lymphoma; Cutaneous B-cell Non-Hodgkin Lymphoma; Extranodal Marginal Zone B-cell Lymphoma of Mucosa-associated Lymphoid Tissue; Hepatosplenic T-cell Lymphoma; Intraocular Lymphoma; Nodal Marginal Zone B-cell Lymphoma; Peripheral T-cell Lymphoma; Recurrent Adult Burkitt Lymphoma; Recurrent Adult Diffuse Large Cell Lymphoma; Recurrent Adult Diffuse Mixed Cell Lymphoma; Recurrent Adult Diffuse Small Cleaved Cell Lymphoma; Recurrent Adult Grade III Lymphomatoid Granulomatosis; Recurrent Adult Immunoblastic Large Cell Lymphoma; Recurrent Adult Lymphoblastic Lymphoma; Recurrent Adult T-cell Leukemia/Lymphoma; Recurrent Colon Cancer; Recurrent Cutaneous T-cell Non-Hodgkin Lymphoma; Recurrent Grade 1 Follicular Lymphoma; Recurrent Grade 2 Follicular Lymphoma; Recurrent Grade 3 Follicular Lymphoma; Recurrent Mantle Cell Lymphoma; Recurrent Marginal Zone Lymphoma; Recurrent Melanoma; Recurrent Mycosis Fungoides/Sezary Syndrome; Recurrent Rectal Cancer; Recurrent Small Lymphocytic Lymphoma; Refractory Hairy Cell Leukemia; Small Intestine Lymphoma; Splenic Marginal Zone Lymphoma; T-cell Large Granular Lymphocyte Leukemia; Testicular Lymphoma; Waldenström Macroglobulinemia
MeSH Terms: conditions — Lymphoma, Extranodal NK-T-Cell; Lymphoma, Large-Cell, Anaplastic; Immunoblastic Lymphadenopathy; Intraocular Lymphoma; Lymphoma, B-Cell, Marginal Zone; Lymphoma, T-Cell, Peripheral; Burkitt Lymphoma; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin; Lymphoma, Large-Cell, Immunoblastic; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Colonic Neoplasms; Lymphoma, T-Cell, Cutaneous; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Melanoma; Mycosis Fungoides; Sezary Syndrome; Rectal Neoplasms; Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia, Hairy Cell; Leukemia, Large Granular Lymphocytic; Waldenstrom Macroglobulinemia | interventions — Ipilimumab; CTLA-4 Antigen; Radiotherapy; Radiation

STUDY DESIGN:
Intervention Model Description: Phase 1 ipilimumab 25 mg safety only. Subsequent Phase 2 ipilimumab 25 mg and radiation combination (treatment-escalation) was not conducted.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ipilimumab 25 mg (Phase 1) (Experimental): Participants receive ipilimumab intratumorally on Day 1
  Interventions: Biological: Ipilimumab
- Ipilimumab 25 mg and radiation therapy (Phase 2) (Experimental): Participants receive ipilimumab intratumorally on Day 1 and undergo local radiation therapy (10 Gy/fraction) within 48 hours for at least 3 fractions
  Interventions: Biological: Ipilimumab; Radiation: Radiation therapy

INTERVENTIONS:
Biological: Ipilimumab — Given intratumorally
  Other Names: Anti-cytotoxic T-lymphocyte-associated antigen-4 monoclonal antibody; MDX-010; MDX-CTLA-4; Monoclonal antibody CTLA-4
Radiation: Radiation therapy — Undergo local radiation therapy, 10 Gy x 3 fractions
  Other Names: Irradiation; Radiotherapy; Therapy, radiation
  Arms: Ipilimumab 25 mg and radiation therapy (Phase 2)

SUMMARY:
This pilot phase 1-2 trial studies the side effects and best of dose ipilimumab when given together with local radiation therapy and to see how well it works in treating patients with recurrent melanoma, non-Hodgkin lymphoma, colon, or rectal cancer. Monoclonal antibodies, such as ipilimumab, can block cancer growth in different ways. Some block the ability of cancer cells to grow and spread. Others find cancer cells and help kill them or carry cancer-killing substances to them. Radiation therapy uses high energy x rays to kill cancer cells. Giving monoclonal antibody therapy together with radiation therapy may be an effective treatment for melanoma, non-Hodgkin lymphoma, colon, or rectal cancer.

* The phase 1 component ("safety") of this study is ipilimumab 25 mg monotherapy.
* The phase 2 component ("treatment-escalation") of this study is ipilimumab 25 mg plus radiation combination therapy.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

1. To assess the safety of combining intratumoral anti-cytotoxic T-lymphocyte-associated protein 4 (CTLA4) immunotherapy with local radiation therapy in patients with melanoma, non-Hodgkin lymphoma, and colorectal carcinoma with a monotherapy ipilimumab safety lead-in.

SECONDARY OBJECTIVES:

1. To assess the induction of an anti-tumor immune responses using laboratory correlative studies.
2. To determine tumor response rates and duration of response at unirradiated tumor sites in patients with advanced malignancies.
3. To identify putative immunologic biomarkers of tumor response.

OUTLINE: This is a phase I safety study of ipilimumab monotherapy, followed by a phase 2 study. Only a few subjects participated in the phase 1 portion of this study. The phase 2 treatment-escalation portion of this study (ipilimumab plus radiation combination therapy) was not conducted.

Patients receive ipilimumab intratumorally on day 1 and undergo local radiation therapy within 48 hours for at least 3 fractions.

After completion of study treatment, patients are followed up at 4 and 8 weeks, and then every 24 weeks for 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to give written informed consent

  * Before any study procedures are performed, subjects (or their legally acceptable representatives) will have the details of the study described to them, and they will be given a written informed consent document to read; then, if subjects consent to participate in the study, they will indicate that consent by signing and dating the informed consent document in the presence of study personnel
* Histologically confirmed malignancy

  * In Phase 1, histologically confirmed melanoma.
  * In Phase 2, histologically confirmed melanoma, non-Hodgkin lymphoma, or colorectal carcinoma
* Must have failed at least 1 systemic therapy or be intolerant to at least one prior systemic treatment
* Must have at least 2 lesions of evaluable size by modified World Health Organization (mWHO)/Cheson criteria; 1 of 2 lesions must be amenable to biopsy (core or fine needle aspirate) and intratumoral injection of up to 5 mL (diameter ≥ 10mm)
* Subjects with asymptomatic brain metastases are eligible; (systemic steroids should be avoided if possible, or the subject should be stable on the lowest clinically effective dose, as steroids as they may interfere with the activity of ipilimumab if administered at the time of the first ipilimumab dose)
* Must be at least 28 days since treatment with standard or investigational chemotherapy, biochemotherapy, surgery, radiation, cytokine therapy, or immunotherapy, and recovered from any clinically significant toxicity experienced during treatment
* Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2
* Life expectancy of ≥ 16 weeks
* Subjects must have baseline (screening/baseline) radiographic images, (e.g. brain, chest, abdomen, pelvis, and bone scans with specific imaging tests to be determined by the attending physician) within 6 weeks of initiation of ipilimumab
* White blood cell (WBC) ≥ 2000/uL (~2 x 10^9/L)
* Absolute neutrophil count (ANC) ≥ 1000/uL (~0.5 x 10^9/L)
* Platelets ≥ 75 x 10^3/uL (~75 x 10^9/L)
* Hemoglobin ≥ 9 g/dL (may be transfused)
* Creatinine ≤ 2.0 x upper limit of normal (ULN)
* Aspartate aminotransferase (AST)/alanine aminotransferase (ALT) ≤ 2.5 x ULN for subjects without liver metastasis ≤ 5 times for liver metastases
* Bilirubin ≤ 2.0 x ULN (except for subjects with Gilbert's syndrome, who must have a total bilirubin of less than 3.0 mg/dL)
* No active or chronic infection with human immunodeficiency virus (HIV), hepatitis B, or hepatitis C
* Women of childbearing potential (WOCBP) must be using an adequate method of contraception to avoid pregnancy throughout the study and for up to 26 weeks after the last dose of investigational product, in such a manner that the risk of pregnancy is minimized; WOCBP include any female who has experienced menarche and who has not undergone successful surgical sterilization (hysterectomy, bilateral tubal ligation, or bilateral oophorectomy) or is not post-menopausal; post-menopause is defined as:

  * Amenorrhea ≥ 12 consecutive months without another cause, or
  * For women with irregular menstrual periods and taking hormone replacement therapy (HRT), a documented serum follicle stimulating hormone (FSH) level ≥ 35 mIU/mL
* Women who are using oral contraceptives, other hormonal contraceptives (vaginal products, skin patches, or implanted or injectable products), or mechanical products such as an intrauterine device or barrier methods (diaphragm, condoms, spermicides) to prevent pregnancy, or are practicing abstinence or where their partner is sterile (eg, vasectomy) should be considered to be of childbearing potential; WOCBP must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of human chorionic gonadotropin [HCG]) within 72 hours before the start of ipilimumab
* Men of fathering potential must be using an adequate method of contraception to avoid conception throughout the study (and for up to 26 weeks after the last dose of investigational product) in such a manner that the risk of pregnancy is minimized

Exclusion Criteria:

* Any other malignancy from which the patient has been disease-free for less than 5 years, with the exception of adequately treated and cured basal or squamous cell skin cancer, superficial bladder cancer or carcinoma in situ of the cervix
* Autoimmune disease: patients with a history of inflammatory bowel disease, including ulcerative colitis and Crohn's disease, are excluded from this study, as are patients with a history of symptomatic disease (eg, rheumatoid arthritis, systemic progressive sclerosis [scleroderma], systemic lupus erythematosus, autoimmune vasculitis [eg, Wegener's Granulomatosis]); motor neuropathy considered of autoimmune origin (e.g. Guillain-Barre Syndrome and Myasthenia Gravis)
* Any underlying medical or psychiatric condition, which in the opinion of the investigator will make the administration of ipilimumab hazardous or obscure the interpretation of adverse events (AEs), such as a condition associated with frequent diarrhea
* Patients with underlying heart conditions who are deemed ineligible for surgery by cardiology consult
* Any non-oncology vaccine therapy used for prevention of infectious diseases (for up to 1 month before or after any dose of ipilimumab)
* A history of prior treatment with ipilimumab or prior CD137 agonist or CTLA 4 inhibitor or agonist
* Concomitant therapy with any of the following: interleukin-2 (IL 2), interferon, or other non-study immunotherapy regimens; cytotoxic chemotherapy; immunosuppressive agents; other investigation therapies; or chronic use of systemic corticosteroids

  * A history of AEs with prior IL-2 or Interferon will not preclude subjects from entering the current study
* Any investigational agents
* Immunosuppressive agents (unless required for treating potential AEs)
* Chronic systemic corticosteroids (unless required for treating treatment emergent AEs or required for management of signs or symptoms due to brain metastases, upon discussion with Bristol-Myers Squibb [BMS] medical monitor)
* Prisoners or subjects who are compulsorily detained (involuntarily incarcerated) for treatment of either a psychiatric or physical (eg, infectious) illness
* Women of childbearing potential (WOCBP) who:

  * Are unwilling or unable to use an acceptable method of contraception to avoid pregnancy for their entire study period and for at least 8 weeks after cessation of study drug, or
  * Have a positive pregnancy test at baseline, or
  * Are pregnant or breastfeeding
* Persons of reproductive potential must agree to use an adequate method of contraception throughout treatment and for at least 8 weeks after ipilimumab is stopped; sexually active WOCBP must use an effective method of birth control during the course of the study, in a manner such that risk of failure is minimized; before study enrollment, WOCBP must be advised of the importance of avoiding pregnancy during study participation and the potential risk factors for an unintentional pregnancy; all WOCBP MUST have a negative pregnancy test before first receiving ipilimumab; if the pregnancy test is positive, the patient must not receive ipilimumab and must not be enrolled in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2013-02; Primary Completion 2014-11 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: George A. Fisher, MD, PhD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Ipilimumab 25 mg: Participants receive ipilimumab intratumorally on Day 1
  Ipilimumab: Given intratumorally
- Ipilimumab 25 mg and Radiation Therapy: Participants receive ipilimumab intratumorally on Day 1 and undergo local radiation therapy (10 Gy/fraction) within 48 hours for at least 3 fractions
  Ipilimumab: Given intratumorally
  Radiation therapy: Undergo local radiation therapy, 10 Gy x 3 fractions
Period: Study Phase 1
Arm/Group | Ipilimumab 25 mg | Ipilimumab 25 mg and Radiation Therapy
Started | 3 | 0
Completed | 3 | 0
Not Completed | 0 | 0
Period: Study Phase 2
Arm/Group | Ipilimumab 25 mg | Ipilimumab 25 mg and Radiation Therapy
Started | 0 | 0
Completed | 0 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ipilimumab 25 mg | Ipilimumab 25 mg and Radiation Therapy | Total
Number analyzed (Participants) | 3 | 0 | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 0 | 2
  >=65 years | 1 | 0 | 1
Age, Continuous [Median (Full Range); unit: years] | 61 [58 to 78] |  | 61 [58 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 |  | 2
  Male | 1 |  | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 |  | 0
  Not Hispanic or Latino | 3 |  | 3
  Unknown or Not Reported | 0 |  | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 |  | 0
  Asian | 0 |  | 0
  Native Hawaiian or Other Pacific Islander | 0 |  | 0
  Black or African American | 0 |  | 0
  White | 3 |  | 3
  More than one race | 0 |  | 0
  Unknown or Not Reported | 0 |  | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 3 |  | 3

OUTCOME MEASURES:

1. Primary Outcome: Dose-limiting Toxicity
Description: Safety as the percentage of patients in Phase 1 (ipilimumab monotherapy) of the study, who experienced dose-limiting toxicities (DLTs) or serious adverse events (SAEs), using National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.0.
Time Frame: 4 weeks
Population: This study did not proceed to Phase 2 (ipilimumab plus radiation combination therapy).
Measure: Number; unit: percentage of participants
Arm/Group | Ipilimumab 25 mg | Ipilimumab 25 mg and Radiation Therapy
Number analyzed (Participants) | 3 | 0
percentage of participants | 0 |

2. Secondary Outcome: Immune Response (Phase 2 Only)
Description: Data will be summarized using proportions with exact 95% confidence intervals, means, standard deviations, and ranges.
Time Frame: 4 weeks
Population: This was a study phase 2 outcome, and no participants were enrolled in study phase 2.
Arm/Group | Ipilimumab 25 mg | Ipilimumab 25 mg and Radiation Therapy
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Immune Response (Phase 2 Only)
Description: Data will be summarized using proportions with exact 95% confidence intervals, means, standard deviations, and ranges.
Time Frame: 8 weeks
Arm/Group | Ipilimumab 25 mg | Ipilimumab 25 mg and Radiation Therapy
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Response Rate (Phase 2 Only)
Description: Response rates calculated based on the Response Evaluation Criteria in Solid Tumors (RECIST)/RECIST Immunotherapy and Cheson criteria (Phase 2 only). Response rate data will be summarized using proportions with exact 95% confidence intervals, means, standard deviations, and ranges.
Time Frame: 8 weeks
Population: This was a study phase 2 outcome, and no participants were enrolled in study phase 2.
Arm/Group | Ipilimumab 25 mg | Ipilimumab 25 mg and Radiation Therapy
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Overall Survival (Phase 2 Only)
Description: Data will be summarized using Kaplan-Meier estimates for time to event data.
Time Frame: Up to 5 years
Population: This was a study phase 2 outcome, and no participants were enrolled in study phase 2.
Arm/Group | Ipilimumab 25 mg | Ipilimumab 25 mg and Radiation Therapy
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Duration of Response (Phase 2 Only)
Description: Data will be summarized using Kaplan-Meier estimates for time to event data.
Time Frame: Up to 5 years
Population: This was a study phase 2 outcome, and no participants were enrolled in study phase 2.
Arm/Group | Ipilimumab 25 mg | Ipilimumab 25 mg and Radiation Therapy
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Ipilimumab 25 mg | Ipilimumab 25 mg and Radiation Therapy
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/0
Other Adverse Events (participants affected / at risk) | 1/3 | 0/0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ipilimumab 25 mg (N=3) | Ipilimumab 25 mg and Radiation Therapy (N=0)
Pain, injection site (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No